CLINICAL TRIAL: NCT06888752
Title: A Clinical Study to Evaluate the Safety, Tolerance and Efficacy of LCAR-M61SQ Cell in Patients with Relapsed/Refractory Multiple Myeloma.
Brief Title: LCAR-M61SQ in Treatment of Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Beijing Boren Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2403-0001
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: multiple myeloma; Relapsed/Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Carboxylesterase

STUDY DESIGN:
Intervention Model Description: Single Group Assignment ，LCAR-61SQ cells intravenous infusion Pretreatment of cyclophosphamide and fludarabine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LCAR-M61SQ (Experimental): Each subject will be given a single-dose LCAR-M61SQ cells infusion at each dose level
  Interventions: Biological: Cell injection

INTERVENTIONS:
Biological: Cell injection — LCAR-M61SQ cells intravenous infusion; Prior to infusion of the LCAR-M61SQ cell, Subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
A prospective, open-label dose-exploration and expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor efficacy characteristics of LCAR-M61SQ in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This study is a prospective, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics, and antitumor efficacy characteristics of LCAR-M61SQ in patients with relapsed/refractory multiple myeloma. All subjects who meet the eligibility criteria will receive intravenous injection of LCAR-M61SQ cell injection. The study will include the following sequential phases: screening, apheresis, pre-treatment (lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in clinical research;
* Age ≥18 years old;
* Eastern Cooperative Oncology Group (ECOG) score 0-2;
* Examination evidence of initial diagnosis of MM according to IMWG diagnostic criteria;
* Measurable lesions were present;
* Subjects have received at least three previous lines of multiple myeloma therapy, each with at least one complete therapy cycle, unless the best response to the therapeutic regimen was documented as disease progression (PD confirmed according to IMWG criteria);
* Expected survival ≥3 months;
* Clinical laboratory values in the screening period meet criteria;

Exclusion Criteria:

* Received previous therapy targeting GPRC5D targets;
* Prior antineoplastic therapy and meet exclusion criteria (before apheresis);
* Subjects had Waldenstrom macroglobulinemia, POEMS syndrome, or primary AL amyloidosis at the time of screening.
* Subjects who were positive for any of HBsAg, HBV DNA, HCV-Ab, HCV RNA, and HIV-Ab;
* Life-threatening allergic reactions, hypersensitivity reactions, or intolerance to CAR-T cell formulations or their excipients, including DMSO, are known.
* Serious underlying diseases were present;
* Female subjects who were pregnant, breastfeeding, or planning to become pregnant while participating in this study or within 1 year of receiving study treatment.
* Also enrolled in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate. | From LCAR-M61SQ cell infusion (Day 1) until the 30th day of follow-up period, assessed up to 30 days
  DLT is classified according to the NCI-CTCAE V5.0 toxicity evaluation criteria and ASTCT consensus classification within 30 days after dose infusion (D1-D30), which is considered by the investigator or collaborator to be reasonably related to LCAR-M61SQ cell therapy.
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | From the date of signing ICF to the date (2 years after LCAR-M61SQcell infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
To determine the recommended dose for phase II clinical trials (RP2D) | through the last subject of DLT exploration completion, about 2years.
  RP2D established through accelerated titration design (ATD) and Bayesian Optimal Interval (BOIN) design.
Maximum concentration (Cmax) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  The maximum observed concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Time to Cmax | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  The time it takes to reach the maximum concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Time to the last observed concentration | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  The time it takes to reach the last observed concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Area Under the Curve (AUC) of the concentration | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  The exposure of CAR positive T cells or transgene CAR copy number in peripheral blood experienced by the subject in a certain time interval.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. ORR is defined as the proportion of patients with PR or better response after infusion of LCAR-M61SQ cells.
Very Good Partial Response Rate（VGPR） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving VGPR according to IMWG criteria.
Complete response（CR） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving CR according to IMWG criteria.
Stringent complete response（sCR） | : From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving sCR according to IMWG criteria.
Minimal residual disease (MRD) negative rate | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression，assessed about 2 years
  Proportion of subjects achieving minimal residual disease (MRD) negative rate according to IMWG criteria.
Time-to-response（TTR） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. TTR is defined as the interval from the date of the first infusion of the LCAR-M61SQ cells to the date of the first efficacy assessment for which the subject met all criteria for PR or better. Analyses were performed only in responders.
Duration of response（DOR） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. DOR is defined as the time from the first documented response (PR or better response) to the first documented evidence of disease progression (as defined according to IMWG criteria) or death from any cause .
Progression-free survival（PFS） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. PFS is defined as the interval from the date of the first infusion of the LCAR-M61SQ cells to the first documentation of disease progression (according to IMWG criteria) or death from any cause, whichever occurred first.
Overall survival（OS | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria.
  Overall survival (OS) is defined as the interval from the date of the first infusion of LCAR-M61SQ cells to death.
Occurrence rate of antidrug antibody | From LCAR-M61SQ cells infusion until the date of first documented progression or study completion，assessed about 2 years
  Occurrence rate of LCAR-M61SQ cells preparation ADA.

IPD SHARING:
Plan to Share IPD: No